CLINICAL TRIAL: NCT05284877
Title: The Organ Transplant Recipient HPV and Skin Cancer Study
Status: Recruiting | Type: Observational
Sponsor: Merete Haedersdal (Other)
Collaborators: Danish Cancer Society (Other); Zealand University Hospital (Other); Vejle Hospital (Other); Herlev and Gentofte Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Merete Haedersdal, Principal investigator, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Other Study IDs: HPV Skin Cancer OTR; Journal-nr.: H-21038387 (Other: National Committee on Health Research Ethics (NVK; Denmark))
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Solid Organ Transplant Recipient; Skin Cancer; Skin Dysplasia; HPV Infection; Cervical Intraepithelial Neoplasia; Cervical Cancer; HPV-Related Malignancy
Keywords: Organ transplant recipient; Skin cancer; Skin dysplasia; Human papillomavirus; HPV-related dysplasia; HPV-related cancer; HPV
MeSH Terms: conditions — Skin Neoplasms; Papillomavirus Infections; Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Whole blood samples from all OTRs at baseline and 6 months after the baseline visit.
  Cervico-vaginal self-sample from all female OTRs and controls at baseline and 12 months after the baseline visit.
  Oral mouthwash sample from all female OTRs and controls at baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Male organ transplant recipients: 300 men with a solid organ transplant (heart, lung, liver, kidney or pancreas)
  Interventions: Other: No intervention
- Female organ transplant recipients: 600 women with a solid organ transplant (heart, lung, liver, kidney or pancreas)
  Interventions: Other: No intervention
- Female immunocompetent controls: 600 immunocompetent women without organ transplant or other immunosuppressive conditions/treatments
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — The study is an observational study without intervention.

SUMMARY:
Solid organ transplant recipients (OTRs) receive lifelong immunosuppressive therapy, which puts them at increased risk of cutaneous and mucosal cancers. In particular, OTRs have increased risk of skin cancer and cancers caused by human papillomavirus (HPV), including cervical cancer and oropharyngeal cancer. There is currently limited knowledge on risk factors for HPV infection and skin cancer in OTRs, and limited knowledge on the natural history of HPV infection and cervical neoplasia in OTRs compared with immunocompetent controls. With a continuously increasing number of OTRs, there is a growing need to improve our understanding of the long-term reactions to immunosuppression.

The overall aim of this study is to investigate long term effects of immunosuppression on cutaneous and mucosal epithelium in Danish OTRs, including the risk of skin dysplasia and skin cancer, cervical and oral HPV infection and HPV-related dysplasia and cancer in OTRs.

This study will be designed as a prospective observational cohort study based on clinical data and data from nationwide Danish registries. A total of 600 female OTRs, 300 male OTRs and 600 female controls will be included from Danish dermatology departments.

The study aims to provide knowledge relevant for improving prevention of skin- and HPV-related cancers in OTRs, including personalized screening recommendations according to individual patient risk.

DETAILED DESCRIPTION:
AIMS

The specific research objectives of this study are:

1. To investigate the overall and type-specific prevalence, incidence and persistence of cervical HPV infection in OTRs compared to immunocompetent controls.
2. To investigate the overall and type-specific prevalence of oral HPV infection in female OTRs compared to immunocompetent controls.
3. To determine the role of lifestyle and clinical factors for the occurrence of cervical and oral HPV infection in female OTRs.
4. To investigate the prevalence and incidence of HPV-related dysplasia and cancer in female OTRs compared with immunocompetent controls.
5. To determine the role of lifestyle, clinical and organ transplantation-related factors for the prevalence and incidence of skin dysplasia in OTRs.
6. To investigate associations between skin dysplasia and prevalence of cervical HPV infection and VZV infection in OTRs.

METHODS

The study will be designed as a clinical prospective cohort study. A total of 600 female OTRs, 300 male OTRs and 600 female immunocompetent controls will be included from the Departments of Dermatology at Bispebjerg, Gentofte and Roskilde Hospitals, Denmark.

The following data will be collected from OTRs:

* At baseline: Questionnaire, dermatologic skin assessment, assessment of skin photodamage (only OTRs recruited from Bispebjerg Hospital), medical record information, cervico-vaginal HPV self-sample test (women only), oral sample for HPV test (women only), blood sample for future research, blood sample for vitamin D test (only OTRs recruited from Bispebjerg Hospital).
* After 6 months: New blood sample for vitamin D test (only OTRs recruited from Bispebjerg Hospital).
* After 12 months: New cervico-vaginal HPV self-sample test (women only).

The following data will be collected from female immunocompetent controls:

* At baseline: Questionnaire, cervico-vaginal HPV self-sample test, oral sample for HPV test.
* After 12 months: New cervico-vaginal HPV self-sample test.

A REDCap database will be established for study data. The RedCap database is encrypted and accessed electronically with personal user-ID and password.

The study population will be linked with nationwide Danish registries and clinical databases. From these registers information on cases of precancerous lesions and cancer; other HPV-related conditions; participation in HPV vaccination and cervical cancer screening; co-morbidities, pregnancies, births and medicine use; socio-demographic characteristics; and emigration and death of women in the study population will be obtained. Registry linkage will be performed for up to 15 years after end of study.

ELIGIBILITY:
Inclusion Criteria for OTRs:

* Patients aged ≥18 years
* Solid organ transplantation recipients, i.e. kidney-, liver-, lung-, and heart transplant recipients
* Stable immunosuppressive treatment for ≥3 months
* No signs of acute graft rejection
* Patients who reside in Denmark
* Informed written consent obtained

Exclusion Criteria for OTRs:

* Patients with concomitant bone marrow transplantation
* Full hysterectomy

Inclusion Criteria for Control group:

* Able patients aged ≥18 years
* No known immunosuppressive therapy or -condition
* Patients who reside in Denmark
* Informed written consent obtained

Exclusion Criteria for Control group:

- Full hysterectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: OTRs attending regular skin cancer screening at the Departments of Dermatology at Bispebjerg Hospital (BBH), Gentofte University Hospital (GEH) and Zealand University Hospital Roskilde (ZUH) are eligible for inclusion in the cohort. Approximately 850 OTR patients are currently attending dermatologic screening at BBH, 400 at GEH, and 450 at ZUH.
  A total of 900 OTRs (300 men and 600 women) will be included. Patient inclusion will be distributed between the three dermatologic departments.
  An immunocompetent control group of women (n=600) will be recruited from the outpatient clinic at the Departments of Dermatology BBH, GEH and ZUH. Controls will be matched with female OTRs according to age (categories 18-29 years, 30-39 years, 40-49 years, 50-59 years, 60-69 years, ≥70 years).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2043-03 (Estimated)

PRIMARY OUTCOMES:
Difference in prevalence, incidence and persistence of cervical HPV infection in female OTRs compared to immunocompetent controls. | Evaluated at baseline and month 12
  Number of women with cervical HPV infection measured by PCR test.

SECONDARY OUTCOMES:
Difference in prevalence of oral HPV infection in female OTRs compared to immunocompetent controls. | Evaluated at baseline
  Number of women with oral HPV infection measured by PCR test.
Correlations between lifestyle factors, clinical factors and occurrence of cervical HPV infection in female OTRs. | Evaluated at baseline
  Lifestyle factors determined by questionnaire. Clinical factors from medical records. Number of women with cervical HPV infection measured by PCR test.
Correlations between lifestyle factors, clinical factors and occurrence of oral HPV infection in female OTRs. | Evaluated at baseline
  Lifestyle factors determined by questionnaire. Clinical factors from medical records. Number of women with oral HPV infection measured by PCR test.
Difference in prevalence and incidence of HPV-related dysplasia and cancer in female OTRs compared to immunocompetent controls. | Evaluated at baseline and during up to 15 years after baseline.
  Number of women with HPV-related dysplasia and HPV-related cancer from registries using registry linkage.
Correlations between lifestyle factors, clinical factors and prevalence of skin dysplasia and cancer in OTRs. | Evaluated at baseline
  Lifestyle factors determined by a questionnaire. Clinical factors from medical records. Skin dysplasia and skin cancer assessed by clinical evaluation and by non-invasive imaging.
Correlation between Vitamin D and prevalence of skin dysplasia and cancer in OTRs. | Evaluated at baseline
  Vitamin D from blood sample analysis. Skin dysplasia and skin cancer assessed by clinical evaluation and non-invasive imaging.
Correlations between skin pigmentation, facial solar lentigines and prevalence of skin dysplasia and cancer in OTRs. | Evaluated at baseline
  Skin pigmentation measured with skin reflectance. Facial solar lentigines measured by photographs. Skin dysplasia and skin cancer assessed by clinical evaluation and non-invasive imaging.
Correlation between prevalence of cervical HPV infection and prevalence of skin dysplasia and cancer in OTRs. | Evaluated at baseline
  Number of women with cervical HPV infection measured by PCR test. Skin dysplasia and skin cancer assessed by clinical evaluation and non-invasive imaging.
Correlations between history of herpes zoster, prevalence of cervical HPV infection and prevalence of skin dysplasia and cancer in OTRs. | Evaluated at baseline
  Number of women with history of herpes zoster determined by questionnaire. Number of women with cervical HPV infection measured by PCR test. Skin dysplasia and skin cancer assessed by clinical evaluation and non-invasive imaging.
Difference in prevalence and incidence of skin cancer in female OTRs compared to immunocompetent controls. | Evaluated at baseline and during up to 15 years after baseline.
  Number of women with skin cancer from registries using registry linkage

CONTACTS AND LOCATIONS:
Overall Officials: Merete Hædersdal, DMSc, MD, Principal Investigator — Bispebjerg Hospital
Locations (3):
- Denmark (3):
  - Department of Dermatology, Bispebjerg Hospital, Copenhagen NV, Capital Region
  - Department of Dermatology and Allergy, Herlev og Gentofte Hospital, Hellerup, Capital Region
  - Department of Dermatology, Zealand University Hospital, Roskilde, Region Sjælland

IPD SHARING:
Plan to Share IPD: Undecided